CLINICAL TRIAL: NCT04537715
Title: A Phase I, Open-label Multi-dose Two-part Study to Characterize the Effects of a Strong CYP3A4 Inhibitor and a Strong CYP3A4 Inducer on the Steady-State Pharmacokinetics of Tazemetostat (EPZ-6438) in Subjects With Advanced Malignancies
Brief Title: Effects of Itraconazole and Rifampin on the Blood Tazemetostat Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EZH-108; 2020-002669-33 (EudraCT Number)
Record Dates: First submitted 2020-07-29; First posted 2020-09-03 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: All Malignancies; Advanced Malignancies; Hematologic Malignancy; Solid Tumor; Follicular Lymphoma (FL); Non-Hodgkin Lymphoma (NHL); Diffuse Large B-Cell Lymphoma (DLBCL); Epithelioid Sarcoma (ES); Synovial Sarcoma; Renal Medullary Carcinoma; Mesothelioma; Rhabdoid Tumor
Keywords: Epizyme; Tazverik; Tazemetostat (EPZ-6438); Itraconazole; CYP3A4 inhibitor; Rifampin; CYP3A4 inducer; Drug-Drug Interaction (DDI); Pharmacokinetics (PK)
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Sarcoma; Sarcoma, Synovial; Mesothelioma; Rhabdoid Tumor | interventions — tazemetostat; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Tazemetostat and Itraconazole Drug Interaction Cycle 1 (Experimental): Participants in Part 1 of the study will receive a single oral, 400 mg dose of tazemetostat on Day 1, 15, and Day 36.
  The study participants will receive tazemetostat (oral 400 mg) tablets to be taken twice daily on Days 3 - 14 and Days 21 - 35. In addition, the participants will receive oral 200 mg itraconazole once daily on Days 18 - 38.
  Study participants may continue tazemetostat from Day 40+ at the recommended therapeutic dose (oral 800 mg twice daily) in 28-day cycles.
  Interventions: Drug: Tazemetostat; Drug: Itraconazole
- Part 2:Tazemetostat and Rifampin Drug Interaction Cycle 1 (Experimental): Participants in Part 2 of the study will receive a single oral, 800 mg dose of tazemetostat on Days 1, 15, and Day 36.
  The study participants will receive tazemetostat (oral 800 mg dose) tablets to be taken twice daily on Days 3 - 14 and Days 17 - 23. In addition, the participants will receive oral 200 mg rifampin once daily on Days 17 - 25.
  Study participants may continue tazemetostat from Day 27+ at the recommended therapeutic dose (oral 800 mg twice daily) in 28-day cycles.
  Interventions: Drug: Tazemetostat; Drug: Rifampin

INTERVENTIONS:
Drug: Tazemetostat — A single, oral, 400 mg dose of tazemetostat on Day 1, Day 15, and Day 36; and tazemetostat (oral 400 mg) tablets twice daily on Days 3 - 14 and Days 21 - 35.
  Other Names: EPZ-6438; Tazverik
  Arms: Part 1: Tazemetostat and Itraconazole Drug Interaction Cycle 1
Drug: Itraconazole — Oral 200 mg itraconazole once daily on Days 18 - 38
  Other Names: Sporanox
  Arms: Part 1: Tazemetostat and Itraconazole Drug Interaction Cycle 1
Drug: Tazemetostat — A single, oral, 800 mg dose of tazemetostat on Days 1, 15, and Day 24 ; and tazemetostat (oral 800 mg) twice daily on Days 3 - 14 and on Days 17 - 23.
  Other Names: EPZ-6438; Tazverik
  Arms: Part 2:Tazemetostat and Rifampin Drug Interaction Cycle 1
Drug: Rifampin — Oral 600 mg rifampin once daily on Days 17 - 25.
  Other Names: RIF; Rifampicin; Rifadin; Rimactane
  Arms: Part 2:Tazemetostat and Rifampin Drug Interaction Cycle 1

SUMMARY:
The participants of this study will have advanced malignancies (also known as advanced cancer). The main aim of this trial will be to study the blood levels (known as pharmacokinetics) of the tazemtostat (the study drug) when administered in combination with another drug.

Part 1 of the study will evaluate the interaction between the drugs tazemetostat and itraconazole.

Part 2 of the study will evaluate the interaction between the drugs tazemetostat and rifampin

For both Parts 1 and 2, safety and the level that effects of the study drug can be tolerated (known as tolerability) will be assessed throughout.

DETAILED DESCRIPTION:
This two-part study is designed to characterize the steady-state PK of oral tazemetostat and its metabolite EPZ 6930 when administered as a single and twice daily dose in subjects with advanced malignancies while taken alone or in combination with either itraconazole or rifampin.

Part 1: tazemetostat and Itraconazole Drug Interaction Part 1 of the study will evaluate the drug-drug interaction between tazemetostat and itraconazole in an open-label, fixed sequential cross over design.

Part 2: tazemetostat and Rifampin Drug Interaction Part 2 of the study will evaluate the drug-drug interaction between tazemetostat and rifampin in an open-label, fixed sequential cross over design.

For both Parts 1 and 2, safety and tolerability will be assessed throughout the subject's participation. Subjects must have an end of study visit after 30 days of the last dose of tazemetostat for safety assessment.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female ≥ 18 years age at the time of consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
3. Has the ability to understand informed consent, and provide signed written informed consent.
4. Life expectancy of > 3 months.
5. Histologically and/or cytologically confirmed advanced metastatic or unresectable solid tumors has progressed after treatment for which there are no standard therapies available OR histologically and/or cytologically confirmed hematologic malignancies that have relapsed, or refractory disease, following at least 2 standard lines of systemic therapy for which there are no standard therapies available.

   Note: Subjects with prior radiotherapy will be included; however, radiotherapy alone will not be considered a separate systemic treatment regimen.
6. Must have evaluable or measurable disease.
7. Has all prior treatment (ie, chemotherapy, immunotherapy, radiotherapy) related clinically significant toxicities resolve to ≤ Grade 1 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0 or are clinically stable and not clinically significant, at time of consent.
8. All subjects must have completed any prior chemotherapy, targeted therapy and major surgery ≥ 28 days before study entry. For daily or weekly chemotherapy without the potential for delayed toxicity, a washout period of 14 days or 5 half-lives, whichever is shorter may be acceptable.
9. Has normal hepatic function (per NCI-ODWG criteria) as well as adequate hematologic (bone marrow [BM] and coagulation factors) and renal function.
10. Able to swallow and retain orally-administered medication and without clinically significant gastrointestinal abnormalities that could alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
11. Females of childbearing potential (FCBP) must have a negative serum pregnancy test and must either practice complete abstinence or agree to use a highly effective method of contraception.
12. Male subjects must have had a successful vasectomy OR must either practice complete abstinence or agree to use a latex or synthetic condom during sexual contact with a female of childbearing potential (FCBP) during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation.

    NOTE: Male subjects must not donate sperm during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation.
13. Has a QT interval corrected by Fridericia's formula (QTcF) ≤450 msec.

EXCLUSION CRITERIA:

1. Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression or primary glioblastoma multiforme.
2. Clinically significant bleeding diathesis or coagulopathy.
3. Known hypersensitivity to any of the components of Tazemetostat, itraconazole, or rifampin.
4. Use of concurrent investigational agent or anticancer therapy.
5. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Have a known active infection with hepatitis B virus (HBV), hepatitis C virus (HCV), AND/OR human T-cell lymphotropic virus 1.
7. Subjects taking medications that are known CYP3A4 inducers or inhibitors (including St. John's Wort).
8. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet and all foods that contain those fruits from 24 hours prior to the first dose of study drug until the last dose of study drug.
9. Any condition or medical problem in addition to the underlying malignancy and organ dysfunction that the Investigator feels would pose unacceptable risk.
10. Has a prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN) or T-cell lymphoblastic lymphoma (T-LBL)/ T-cell acute lymphoblastic leukemia (T-ALL).
11. Ingestion of alcohol within 72 hours prior to day 1 of Cycle 1 until the end of Cycle 1 (Day 39 for Part 1 and Day 26 for Part 2). Regular alcohol consumption must not exceed 16 units for males and 7 units for females per week (2 units equals 40mL [a can] of beer, 175mL [a standard glass] of wine, or 50 mL [2 small shots] of spirits
12. Any form of marijuana use.
13. History of drug abuse (including alcohol) within the last 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipse Medical Director, Study Director — Ipsen
Locations (10):
- United States (7):
  - California Cancer Associates for Research and Excellence, Inc. (cCARE), Encinitas, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Northwestern University-Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
- Spain (3):
  - Onkologikoa, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2024/03/28163657/EZH-108-lay-results-summary.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1, 2-part, multi-dose, open-label study was conducted in participants with advanced malignancies from 23 April 2020 to 03 April 2023 at 10 investigational sites in Spain and USA. Part 1 evaluated drug-drug interaction (DDI) between tazemetostat and itraconazole; Part 2 evaluated DDI between tazemetostat and rifampin.
Pre-assignment Details: This study consisted of a screening period (up to 30 days), Part 1 consisted of Cycle 1 till Day 39, Cycle 2 started on Day 40 and each subsequent cycle was of 28-day duration; Part 2 also consisted of Cycle 1 till Day 26, Cycle 2 started on Day 27 of and each subsequent cycle was of 28-day duration until Investigator assessed clinical progression per standard practice, unacceptable treatment related toxicity/withdrawal; survival follow-up (until death/study closure).
Groups:
- Part 1: Tazemetostat + Itraconazole: Participants received a single oral dose of 400 milligram (mg) tazemetostat on Cycle 1 Day 1, twice daily (BID) dose of tazemetostat 400 mg on Days 3 to 14 and single dose of tazemetostat 400 mg on Day 15. A single oral dose of 200 mg itraconazole was administered daily from Day 18 to Day 20. From Days 21 to 35, they received a 400 mg BID dose of tazemetostat co-administered with a single dose of oral 200 mg itraconazole. Itraconazole was also administered on Days 37 and 38 as a single oral 200 mg daily dose. On Cycle 1 Day 36, they received a single dose of 400 mg tazemetostat co-administered with a single dose of oral 200 mg itraconazole. Participants continued to receive tazemetostat treatment at the recommended therapeutic dose (oral 800 mg tazemetostat BID), from Day 40 (Cycle 2 Day 1) for each subsequent cycle of 28-day duration until Investigator assessed clinical progression per standard practice, unacceptable treatment related toxicity/withdrawal; survival follow-up (until death/study closure).
- Part 2: Tazemetostat + Rifampin: Participants received a single oral dose of 800 mg tazemetostat on Cycle 1 Day 1, BID dose of 800 mg of tazemetostat from Days 3 to 14 and a single oral dose of 800 mg tazemetostat on Day 15. From Days 17 to 23, they received an 800 mg BID dose of tazemetostat co-administered with a single dose of oral 600 mg rifampin. On Day 24, subjects received a single dose of 800 mg tazemetostat co-administered with a single dose of oral 600 mg rifampin. Rifampin was also administered on Cycle 1 Day 25 as a single oral 600 mg dose. Participants continued to receive tazemetostat treatment at the recommended therapeutic dose (oral 800 mg tazemetostat BID), from Day 27 (Cycle 2 Day 1) for each subsequent cycle of 28-day duration until Investigator assessed clinical progression per standard practice, unacceptable treatment related toxicity/withdrawal; survival follow-up (until death/study closure).
Period: Overall Study
Arm/Group | Part 1: Tazemetostat + Itraconazole | Part 2: Tazemetostat + Rifampin
Started | 21 | 21
Completed | 10 | 16
Not Completed | 11 | 5
Not completed — Death | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Other | 4 | 3
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Enrolled population included all participants who signed informed consent and met all screening criteria.
Groups:
- Part 1: Tazemetostat + Itraconazole: Participants received a single oral dose of 400 mg tazemetostat on Cycle 1 Day 1, BID dose of tazemetostat 400 mg on Days 3 to 14 and single dose of tazemetostat 400 mg on Day 15. A single oral dose of 200 mg itraconazole was administered daily from Day 18 to Day 20. From Days 21 to 35, they received a 400 mg BID dose of tazemetostat co-administered with a single dose of oral 200 mg itraconazole. Itraconazole was also administered on Days 37 and 38 as a single oral 200 mg daily dose. On Cycle 1 Day 36, they received a single dose of 400 mg tazemetostat co-administered with a single dose of oral 200 mg itraconazole. Participants continued to receive tazemetostat treatment at the recommended therapeutic dose (oral 800 mg tazemetostat BID), from Day 40 (Cycle 2 Day 1) for each subsequent cycle of 28-day duration until Investigator assessed clinical progression per standard practice, unacceptable treatment related toxicity/withdrawal; survival follow-up (until death/study closure).
- Total: Total of all reporting groups
Arm/Group | Part 1: Tazemetostat + Itraconazole | Part 2: Tazemetostat + Rifampin | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.45) | 60.1 (13.05) | 60.5 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 12 | 30
  Asian | 2 | 3 | 5
  Black or African American | 0 | 2 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Not reported/Other | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time 0 to 12 Hours of Quantifiable Concentration (AUC0-12h) of Tazemetostat
Description: Blood samples were collected at specified timepoints. AUC0-12h was assessed using non-compartmental data analysis method. AUC0-12h was estimated by a combination of linear trapezoidal method on concentrations going up and logarithmic trapezoidal method on concentrations going down (Linear up/Log down method).
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: The Pharmacokinetic (PK) population included all participants who had sufficient PK concentration data to calculate steady-state PK parameters in Part 1 and did not have any major protocol deviation that was deemed to greatly alter the steady-state exposure to tazemetostat or itraconazole.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram/milliliter (h*ng/mL)
Groups:
- Part 1: Tazemetostat: Participants received a single oral dose of 400 mg tazemetostat on Cycle 1 Day 1, BID dose of tazemetostat 400 mg on Days 3 to 14 and single dose of tazemetostat 400 mg on Day 15. From Days 21 to 35, they received a 400 mg BID dose of tazemetostat. On Cycle 1 Day 36, they received a single dose of 400 mg tazemetostat. Participants continued to receive tazemetostat treatment at the recommended therapeutic dose (oral 800 mg tazemetostat BID), from Day 40 (Cycle 2 Day 1) for each subsequent cycle of 28-day duration until Investigator assessed clinical progression per standard practice, unacceptable treatment related toxicity/withdrawal; survival follow-up (until death/study closure).
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
hours*nanogram/milliliter (h*ng/mL)
  Cycle 1 Day 1 | 2180 (55.3)
  Cycle 1 Day 15 | 1830 (37.6)

2. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Tazemetostat
Description: Blood samples were collected at specified timepoints. Cmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, 48, and 72 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: The PK population included all participants who had sufficient PK concentration data to calculate steady-state PK parameters in Part 1 and did not have any major protocol deviation that was deemed to greatly alter the steady-state exposure to tazemetostat or itraconazole.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
ng/mL
  Cycle 1 Day 1 | 704 (56.5)
  Cycle 1 Day 15 | 543 (63.3)

3. Primary Outcome: Part 2: AUC0-12h of Tazemetostat
Description: as for outcome 1
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: The PK population included all participants who had sufficient PK concentration data to calculate steady-state PK parameters in Part 2 and did not have any major protocol deviation that was deemed to greatly alter the steady-state exposure to tazemetostat or rifampin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Part 2: Tazemetostat: Participants received a single oral dose of 800 mg tazemetostat on Cycle 1 Day 1, BID dose of 800 mg of tazemetostat from Days 3 to 14 and a single oral dose of 800 mg tazemetostat on Day 15. From Days 17 to 23, they received an 800 mg BID dose of tazemetostat. On Day 24, subjects received a single dose of 800 mg tazemetostat. Participants continued to receive tazemetostat treatment at the recommended therapeutic dose (oral 800 mg tazemetostat BID), from Day 27 (Cycle 2 Day 1) for each subsequent cycle of 28-day duration until Investigator assessed clinical progression per standard practice, unacceptable treatment related toxicity/withdrawal; survival follow-up (until death/study closure).
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
h*ng/mL
  Cycle 1 Day 1 | 4420 (83.2)
  Cycle 1 Day 15 | 3610 (70.3)

4. Primary Outcome: Part 2: Cmax of Tazemetostat
Description: Blood samples were collected at specified timepoints. Cmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
ng/mL
  Cycle 1 Day 1 | 1330 (67.4)
  Cycle 1 Day 15 | 1100 (78.7)

5. Secondary Outcome: Part 1: AUC0-12h of EPZ-6930 After Tazemetostat Alone at Steady-State
Description: as for outcome 1
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose on Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
h*ng/mL | 3650 (26.4)

6. Secondary Outcome: Part 1: AUC0-12h of Tazemetostat and EPZ-6930 After Tazemetostat at Steady-State With Itraconazole
Description: as for outcome 1
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose on Cycle 1 Day 36
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
h*ng/mL
  Tazemetostat | 4530 (64.5)
  EPZ-6930 | 5450 (46.6)

7. Secondary Outcome: Part 1: Cmax of EPZ-6930 After Tazemetostat Alone at Steady-State
Description: Blood samples were collected at specified timepoints. Cmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
ng/mL | 780 (38.2)

8. Secondary Outcome: Part 1: Cmax of Tazemetostat and EPZ-6930 After Tazemetostat at Steady State With Itraconazole
Description: Blood samples were collected at specified timepoints. Cmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 36
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
ng/mL
  Tazemetostat | 1010 (76.3)
  EPZ-6930 | 792 (44.7)

9. Secondary Outcome: Part 1: Observed Time at Cmax (Tmax) of Tazemetostat and EPZ-6930 After Tazemetostat Alone at Steady-State
Description: Blood samples were collected at specified timepoints. Tmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
hour
  Tazemetostat | 1.34 (72.1)
  EPZ-6930 | 1.70 (51.4)

10. Secondary Outcome: Part 1: Tmax of Tazemetostat and EPZ-6930 After Tazemetostat at Steady-State With Itraconazole
Description: Blood samples were collected at specified timepoints. Tmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 36
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
hour
  Tazemetostat | 1.55 (63.4)
  EPZ-6930 | 1.82 (49.9)

11. Secondary Outcome: Part 1: Apparent Terminal Elimination Half-Life (t1/2) of Tazemetostat and EPZ-6930 After Tazemetostat Alone at Steady-State
Description: Blood samples were collected at specified timepoints. T1/2 was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 15
Population: The PK population included all participants who had sufficient PK concentration data to calculate steady-state PK parameters in Part 1 and did not have any major protocol deviation that was deemed to greatly alter the steady-state exposure to tazemetostat or itraconazole. Only data from the participants analyzed were reported.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
hour
  Tazemetostat: number analyzed (Participants) | 15
  Tazemetostat | 8.21 [4.67 to 19.8]
  EPZ-6930 | 15.8 [8.10 to 22.8]

12. Secondary Outcome: Part 1: T1/2 of Tazemetostat and EPZ-6930 After Tazemetostat at Steady-State With Itraconazole
Description: Blood samples were collected at specified timepoints. T1/2 was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 36
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
hour
  Tazemetostat: number analyzed (Participants) | 15
  Tazemetostat | 12.8 [6.40 to 22.0]
  EPZ-6930 | 13.9 [7.19 to 21.6]

13. Secondary Outcome: Part 2: AUC0-12h of EPZ-6930 After Tazemetostat Alone at Steady-State
Description: as for outcome 1
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose on Cycle 1 Day 15
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
h*ng/mL | 7010 (72.0)

14. Secondary Outcome: Part 2: AUC0-12h of Tazemetostat and EPZ-6930 After Tazemetostat at Steady-State With Rifampin
Description: as for outcome 1
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose on Cycle 1 Day 24
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2: Tazemetostat + Rifampin
Number analyzed (Participants) | 16
h*ng/mL
  Tazemetostat | 588 (65.2)
  EPZ-6930 | 3070 (34.1)

15. Secondary Outcome: Part 2: Cmax of EPZ-6930 After Tazemetostat Alone at Steady-State
Description: Blood samples were collected at specified timepoints. Cmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose on Cycle 1 Day 15
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
ng/mL | 1530 (49.5)

16. Secondary Outcome: Part 2: Cmax of Tazemetostat and EPZ-6930 After Tazemetostat at Steady State With Rifampin
Description: Blood samples were collected at specified timepoints. Cmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 hours post-dose on Cycle 1 Day 24
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Tazemetostat + Rifampin
Number analyzed (Participants) | 16
ng/mL
  Tazemetostat | 181 (71.7)
  EPZ-6930 | 857 (40.5)

17. Secondary Outcome: Part 2: Tmax of Tazemetostat and EPZ-6930 After Tazemetostat Alone at Steady-State
Description: Blood samples were collected at specified timepoints. Tmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose on Cycle 1 Day 15
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
hour
  Tazemetostat | 1.25 (47.0)
  EPZ-6930 | 1.47 (59.1)

18. Secondary Outcome: Part 2: Tmax of Tazemetostat and EPZ-6930 After Tazemetostat at Steady-State With Rifampin
Description: Blood samples were collected at specified timepoints. Tmax was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 hours post-dose on Cycle 1 Day 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 2: Tazemetostat + Rifampin
Number analyzed (Participants) | 16
hour
  Tazemetostat | 1.40 (1.10)
  EPZ-6930 | 1.85 (0.934)

19. Secondary Outcome: Part 2: T1/2 of Tazemetostat and EPZ-6930 EPZ-6930 After Tazemetostat Alone at Steady-State
Description: Blood samples were collected at specified timepoints. T1/2 was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose on Cycle 1 Day 15
Population: The PK population included all participants who had sufficient PK concentration data to calculate steady-state PK parameters in Part 2 and did not have any major protocol deviation that was deemed to greatly alter the steady-state exposure to tazemetostat or rifampin. Only data from the participants analyzed were reported.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
hour
  Tazemetostat: number analyzed (Participants) | 15
  Tazemetostat | 7.21 [5.55 to 10.6]
  EPZ-6930 | 8.38 [6.44 to 13.8]

20. Secondary Outcome: Part 2: T1/2 of Tazemetostat and EPZ-6930 After Tazemetostat at Steady-State With Rifampin
Description: Blood samples were collected at specified timepoints. T1/2 was assessed using non-compartmental data analysis method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 hours post-dose on Cycle 1 Day 24
Population: as for outcome 19
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: Tazemetostat + Rifampin
Number analyzed (Participants) | 15
hour
  Tazemetostat | 5.24 [2.45 to 8.19]
  EPZ-6930 | 8.07 [3.70 to 10.3]

21. Other Pre Specified Outcome: Part 1: Least Squares Geometric Mean Ratio of Observed Accumulation Ratio of AUC0-12h for Tazemetostat
Description: Blood samples were collected at specified timepoints. AUC0-12h accumulation ratio was assessed using non-compartmental data analysis method. AUC0-12h accumulation ratio was calculated as the ratio of AUC0-12h at steady state (Cycle 1 Day 15) divided by AUC0-12 during the initial dosing interval (Cycle 1 Day 1).
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
ratio | 0.842 [0.726 to 0.976]

22. Other Pre Specified Outcome: Part 1: Least Squares Geometric Mean Ratio of Cmax Accumulation Ratio for Tazemetostat
Description: Blood samples were collected at specified timepoints. Cmax accumulation ratio was assessed using non-compartmental data analysis method. Cmax accumulation ratio was calculated as the ratio of Cmax at steady state (Cycle 1 Day 15) divided by Cmax during the initial dosing interval (Cycle 1 Day 1).
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8,12, 36, 48 post-dose on Cycle 1 Day 1, and 72 hours post-dose on Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 1: Tazemetostat
Number analyzed (Participants) | 16
ratio | 0.771 [0.662 to 0.897]

23. Other Pre Specified Outcome: Part 1: Least Squares Geometric Mean Ratio of AUC0-12h After Single Dose of Tazemetostat With Itraconazole
Description: Blood samples were collected at specified timepoints. Drug-drug interaction was assessed using analysis of variance (ANOVA).
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose on Cycle 1 Day 1 (without itraconazole) and Cycle 1 Day 21 (with itraconazole)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
ratio | 3.12 [2.44 to 3.99]

24. Other Pre Specified Outcome: Part 1: Least Squares Geometric Mean Ratio of Cmax After Single Dose of Tazemetostat With Itraconazole
Description: Blood samples were collected at specified timepoints. Drug-drug interaction was assessed using ANOVA.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose on Cycle 1 Day 1 (without itraconazole) and Cycle 1 Day 21 (with itraconazole)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
ratio | 2.00 [1.60 to 2.48]

25. Other Pre Specified Outcome: Part 1: Least Squares Geometric Mean Ratio of AUC0-12h After Tazemetostat at Steady-State With Itraconazole
Description: Blood samples were collected at specified timepoints. Drug-drug interaction was assessed using ANOVA.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose on Cycle 1 Day 15 (without itraconazole) and Cycle 1 Day 36 (with itraconazole)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
ratio | 2.47 [2.02 to 3.02]

26. Other Pre Specified Outcome: Part 1: Least Squares Geometric Mean Ratio of Cmax After Tazemetostat at Steady-State With Itraconazole
Description: Blood samples were collected at specified timepoints. Drug-drug interaction was assessed using ANOVA.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 36, and 72 hours post-dose on Cycle 1 Day 15 (without itraconazole) and Cycle 1 Day 36 (with itraconazole)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 1: Tazemetostat + Itraconazole
Number analyzed (Participants) | 16
ratio | 1.86 [1.49 to 2.31]

27. Other Pre Specified Outcome: Part 2: Least Squares Geometric Mean Ratio of Observed Accumulation Ratio of AUC0-12h for Tazemetostat
Description: Blood samples were collected at specified timepoints. AUC0-12h accumulation ratio was assessed using non-compartmental data analysis method. AUC0-12h accumulation ratio was calculated as the ratio of AUC0-12h at steady state (Cycle 1 Day 15) divided by AUC0-12h during the initial dosing interval (Cycle 1 Day 1).
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8,12, 24, 36, and 48 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 3
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
ratio | 0.816 [0.638 to 1.04]

28. Other Pre Specified Outcome: Part 2: Least Squares Geometric Mean Ratio of Cmax Accumulation Ratio for Tazemetostat
Description: as for outcome 22
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8,12, 24, 36, and 48 hours post-dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 3
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 2: Tazemetostat
Number analyzed (Participants) | 16
ratio | 0.828 [0.635 to 1.08]

29. Other Pre Specified Outcome: Part 2: Least Squares Geometric Mean Ratio of AUC0-12h After Tazemetostat at Steady State With Rifampin
Description: Blood samples were collected at specified timepoints. Drug-drug interaction was assessed using ANOVA.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose on Cycle 1 Day 15 (without rifampin) and Cycle 1 Day 24 (with rifampin)
Population: as for outcome 3
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 2: Tazemetostat + Rifampin
Number analyzed (Participants) | 16
ratio | 0.163 [0.128 to 0.208]

30. Other Pre Specified Outcome: Part 2: Least Squares Geometric Mean Ratio of Cmax After Tazemetostat at Steady State With Rifampin
Description: Blood samples were collected at specified timepoints. Drug-drug interaction was assessed using ANOVA.
Time Frame: Pre-dose (0 hour), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose on Cycle 1 Day 15 (without rifampin) and Cycle 1 Day 24 (with rifampin)
Population: as for outcome 3
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Part 2: Tazemetostat + Rifampin
Number analyzed (Participants) | 16
ratio | 0.164 [0.122 to 0.219]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events and all-cause mortality were reported from the first dose of study treatment (Day 1) through 30 days after the end of study treatment (approximately 33 months).
Description: The Safety population included all participants in the Enrolled population who received at least 1 dose or partial dose of the study treatments and had 1 post-dose safety observation recorded.
Arm/Group | Part 1: Tazemetostat + Itraconazole | Part 2: Tazemetostat + Rifampin
All-Cause Mortality (participants affected / at risk) | 10/21 | 3/21
Serious Adverse Events (participants affected / at risk) | 8/21 | 9/21
Other Adverse Events (participants affected / at risk) | 19/21 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tazemetostat + Itraconazole (N=21) | Part 2: Tazemetostat + Rifampin (N=21)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Tazemetostat + Itraconazole (N=21) | Part 2: Tazemetostat + Rifampin (N=21)
Anaemia (Blood and lymphatic system disorders) | 6 (10) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (9) | 5 (6)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (6) | 9 (10)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 2 (2)
Asthenia (General disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 4 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04537715/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT04537715/SAP_001.pdf